CLINICAL TRIAL: NCT01305369
Title: The Effect of Prasugrel on Bronchial Hyperreactivity and on Markers of Inflammation in Patients With Chronic Asthma: a Pilot Randomised Controlled Trial (PRINA Study)
Brief Title: The Effect of Prasugrel on Bronchial Hyperreactivity and on Markers of Inflammation in Patients With Chronic Asthma
Acronym: PRINA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Milan (Other)
Responsible Party: Principal Investigator, Marco Cattaneo, Professor, University of Milan
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Prina01
Record Dates: First submitted 2011-02-25; First posted 2011-02-28 (Estimated); Last update posted 2012-03-06 (Estimated); Status verified 2012-03

CONDITIONS: Chronic Asthma
Keywords: ASTHMA; PLATELET RECEPTOR P2Y12; PRASUGREL; INFLAMMATION
MeSH Terms: conditions — Asthma; Inflammation | interventions — Prasugrel Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Prasugrel — Patients will be blindly and randomly allocated to treatment A (prasugrel 10 mg daily) or B (placebo) for 15 days. After a 15-day wash-out period, patients who had initially been allocated to treatment "A" will be allocated to treatment "B", and vice versa.

SUMMARY:
Cysteinyl leukotrienes (cys-LTs) are lipid inflammatory mediators that abound in mucosal inflammation and play a validated role in the pathogenesis of human asthma. It has recently been demonstrated that the platelet adenosine diphosphate (ADP) receptor, P2Y12, is required for LT4-mediated pulmonary inflammation and could be a novel potential therapeutic target for asthma. Thienopyridines (such as ticlopidine and clopidogrel) are pro-drugs, with proven antithrombotic efficacy, whose active metabolites selectively inhibit the platelet P2Y12 receptors. One of the drawbacks of thienopyridines is the high inter-individual variability in pharmacological response, mostly due to the high inter-individual variability in the capacity of transforming the pro-drug in its active metabolite. Prasugrel is a new member of the class of thienopyridines, with faster onset of action and a more uniform inhibition of platelet function compared to the other thienopyridines. Primary objective of our study will be to test whether or not the inhibition of the platelet P2Y12 receptor by prasugrel reduces the bronchial hyper-reactivity in patients with chronic asthma. The investigators designed a randomized, double blind (Subject, Caregiver, Investigator, Outcomes Assessor), crossover, placebo-controlled, prospective study, which will enroll 26 patients. Randomization will be performed in sequential blocks. Patients will be blindly and randomly allocated to treatment A (prasugrel 10 mg daily) or B (placebo) for 15 days. After a 15-day wash-out period, patients who had initially been allocated to treatment "A" will be allocated to treatment "B", and vice versa. Measurements will be done at baseline and on day 15 after each treatment, at the same time (+/- 1 h) of the day. Primary efficacy measure will be changes in airway hyper-responsiveness, recorded as reduction of FEV1 using the mannitol test induction. Secondary efficacy measures will be changes in markers of airway inflammation in sputum, changes in measurement of nitric oxide expiration (as surrogate marker of airway lung inflammation), count of eosinophil granulocytes in peripheral blood smear, changes in asthma exacerbation rates and symptom scores. Changes in phosphorylation of platelet VASP (Vasodilator-stimulated phosphoprotein) by ADP, measured with a flow cytometric technique, will be used as markers of the degree of inhibition of platelet P2Y12 receptors attained in each subjects by treatment with prasugrel.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic asthma, diagnosed based on the occurrence of episodic wheezing, chest tightness and/or dyspnoea and objectively confirmed according to standard criteria, such as methacholine airway hyper-responsiveness (PC20 FEV1 < 16mg/ml) and positivity of skin test to common allergens (prick test)
* Positivity of bronchial challenge testing with mannitol
* Age range of 18-74 years old
* Duration of asthma > 1 year
* Mild and stable asthma without chronic medication, except for the use of inhaled low dose of steroids or the use of inhaled beta2-agonist on demand
* Written informed consent

Exclusion Criteria:

* Pregnancy/lactation
* Active bleeding or high risk of bleeding contraindicating treatment with antiplatelet agents or anticoagulants
* Previous TIA or stroke
* Age ≥ 75 years old
* Other indication for anti-platelet therapy
* Systolic blood pressure > 180 mmHg or diastolic blood pressure > 110 mmHg
* Body weight < 60 Kg
* Use of any FANS in the last 7 days

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2011-03; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Changes in airway hyper-responsiveness | baseline and day 15 after each treatment
  Changes in airway hyper-responsiveness, recorded as reduction of FEV1 with the mannitol test induction. Mannitol is considered more specific respect to methacholine for detecting changes in airway hyper-responsiveness in asthma patients, because it mimics the normal pathophysiology of bronchial asthma, causing the release of various mediators of bronchoconstriction

SECONDARY OUTCOMES:
Changes in measurement of airway inflammation in sputum | At baseline and on day 15 after each treatment
Changes in measurement of nitric oxide expiration | At at baseline and on day 15 after each treatment
  Changes in measurement of nitric oxide expiration, as a surrogate marker of airway lung inflammation
Changes in phosphorylation of platelet VASP | At baseline and on day 15 after each treatment
  Changes in phosphorylation of platelet VASP (Vasodilator-stimulated phosphoprotein) by ADP, measured with a flow cytometric technique, as markers of the degree of inhibition of platelet P2Y12 receptors attained in each subjects by treatment with prasugrel

CONTACTS AND LOCATIONS:
Overall Officials: Marco Cattaneo, MD, Principal Investigator — University of Milan
Locations (1):
- Medicina 3 Ospedale San Paolo Dipartimento di Medicina Chirurgia e Odontoiatria, Università di Milano, Milan, Italy